CLINICAL TRIAL: NCT06443216
Title: Auditory Closed-loop Modulation of Slow Wave Sleep to Treat Major Depressive Disorder
Brief Title: Sleep Modulation to Treat Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christoph Nissen (Other)
Responsible Party: Sponsor-Investigator, Christoph Nissen, Prof. Dr. med., University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2023-01804
Record Dates: First submitted 2024-05-22; First posted 2024-06-05 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Major Depressive Disorder; Healthy
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients with major depressive disorder according to ICD-10 criteria
  Interventions: Device: Auditory closed-loop stimulation; Device: Sham stimulation
- Healthy Group (Experimental): Healthy controls
  Interventions: Device: Auditory closed-loop stimulation; Device: Sham stimulation

INTERVENTIONS:
Device: Auditory closed-loop stimulation — Auditory closed-loop suppression of slow wave sleep
Device: Sham stimulation — No auditory stimulation

SUMMARY:
Current first-line treatments for major depression (antidepressants and psychotherapy) show a long latency to response, and less than half of all patients experience full remission with optimized treatment, indicating the need for new developments. The aim of this study is to extend and further develop a longstanding line of research of using sleep neurophysiology as a 'window to the brain' and treatment development in major depression. Particularly, this project is designed to test the feasibility, efficacy and mechanisms of action of a new sleep-based treatment technology.

DETAILED DESCRIPTION:
The planned study is a single-centre, doubled-blind, randomized, sham controlled, repeated measures within-subject (stimulation and sham) study including patients with major depression and healthy controls, across four sleep laboratory nights (adaptation, baseline, stimulation and sham in counterbalanced order). The investigators will test the primary hypothesis that auditory-closed loop suppression of slow wave sleep will improve depressive clinical symptomatology compared to sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* MDD according to ICD-10 criteria (F32.1/2, F33.1/2; i.e. unipolar depression) for patient group

Exclusion Criteria:

* Relevant psychiatric disorders (other than MDD for the patient group), such as organic psychiatric disorders, lifetime history of substance dependency or current substance abuse (smoking will be allowed for recruitment reasons), schizophrenia or other psychotic disorders, affective disorders including bipolar disorder, borderline personality disorder, autism or other severe psychiatric disorders
* Known pregnancy
* Unstable medical conditions, such as unstable cardiovascular or metabolic disorders, etc.
* Relevant neurological disorders, including epilepsy, stroke, etc.
* Organic sleep disorders including relevant sleep apnea (AHI>15/h), periodic limb movement disorder (PLMS index>5/h), Restless-Legs-Syndrome (RLS), narcolepsy, circadian rhythm disorder or shift work/ jet lag
* Intake of medication affecting the central nervous system (other than antidepressants and lithium in patients); patients receiving benzodiazepines or (es)ketamine will not be included
* Current brain stimulation treatment, such as electroconvulsive therapy (ECT), TMS or deep brain stimulation
* Contraindications for tDCS or TMS studies, including but not limited to metal in the head/ brain or epilepsy
* Hearing impairment or tinnitus (auditory stimulation study)
* Inability to follow the procedures of the study (for example due to language problems)
* Left-handedness

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale | Up to three weeks
  Measure of the severity of depressive symptomatology
  The scores range between 0 to 60. The higher the score, the more symptamology of depression the subjects presents.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Geneva, Geneva, Switzerland